CLINICAL TRIAL: NCT03696940
Title: Estudio clínico Fase III Para Evaluar la Eficacia terapéutica en Pacientes Mexicanos Con Dislipidemia Mediante el Uso vía Oral de L-Carnitina + Atorvastatina Comparado Con Atorvastatina
Brief Title: Clinical Trial to Evaluate the Efficacy of a Dyslipidemic Therapy in Mexican Population
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratorios Grossman, S.A. (Industry)
Collaborators: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMX-001-2017
Record Dates: First submitted 2018-09-18; First posted 2018-10-05 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Dyslipidemias; Cardiovascular Risk Factor
MeSH Terms: conditions — Dyslipidemias | interventions — Carnitine; Tablets; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Longitudinal
Who Masked: Participant
Masking Description: Simple Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 2 tablets of: L-Carnitine 500Mg Oral Tablet + Atorvastatin 10 mg
  Interventions: Drug: L-Carnitine 500Mg Oral Tablet + Atorvastatin 10 mg
- Control Group (Active Comparator): 2 tablets of: Atorvastatin 10 mg
  Interventions: Drug: Atorvastatin 10mg

INTERVENTIONS:
Drug: L-Carnitine 500Mg Oral Tablet + Atorvastatin 10 mg — Oral administration of 2 tablets of atorvastatin 10 mg (each one) every 24 hours for 6 months.
  Other Names: Experimental Group
  Arms: Experimental Group
Drug: Atorvastatin 10mg — Oral administration of 2 tablets atorvastatin 10 mg (each one) every 24 hours for 6 months.
  Other Names: Active control group
  Arms: Control Group

SUMMARY:
Clinical Trial Phase III, experimental, simple blind, randomized with two treatment groups, multicentric, longitudinal, to evaluate the therapuetic efficacy to dislipydemias in mexican adult population. This trial includes homogeneus populations that could be comparable by their disease condition, biologic characteristics and sociodemographics characteristics.

2 Treatment groups: Experimental Group: Oral Administration of L-carnitine (1g) + Oral Atorvastatin (20mg), every 24 hours for 6 months.

Active control group: Oral Administration of Atorvastatin 20mg every 24 hours for 6 months.

Sample Size: 120 subjects, females or males between 35 to 75 years old. Laboratory tests: Hematic biometry, quimical blood components, electrocardiogram and pregnancy urinary test.

DETAILED DESCRIPTION:
General objectives:

Evaluate the therapeutic efficacy in Mexican adults with dyslipidemia through the oral route use of L-carnitine + atorvastatin in comparison with the use of Atorvastatin, after six months of treatment.

Evaluate the safety of the medicines under study.

Hypothesis:

The combined use of L-carnitine + atorvastatin offers therapeutic superiority with respect to the use of atorvastatin as treatment to reduce the percentage of C-LDL in patients with dyslipidemia.

The combination of L-carnitine + atorvastatin shows fewer incidences in the presence of adverse events attributable to the medicine in comparison to the use of atorvastatin as mono-therapy, in the treatment of dyslipidemia patients.

Design:

Phase III clinical assay, experimental randomized with two treatment, multi-centered, longitudinal, to evaluate the therapeutic efficacy in dyslipidemias of Mexican adults.

Material and Methods:

Sample Size 120 subjects will be included. Inclusion Criteria Mexicans between 35 and 75 years of age. Gender indistinct. Patient with abnormal lipid profile considered as serum levels of C-LDL of 100mg/dl or greater obtained by laboratory parameters.

Not under pharmacologic treatment to handle their dyslipidemia or accepting to suspend their current treatment and be evaluated for their inclusion in the next 3 weeks starting on the day of the initial evaluation.

Women in fertile stage with a safe, hormonal-free family planning method. A safe planning method includes surgical methods in women, intrauterine device that doesn't release progestines and use of preservative in all their sexual relations.

Women in fertile stage who don't wish to become pregnant during their participation in the study.

Post-menopause women or with hysterectomy history. Have a fixed and/or mobile telephone and accept to receive calls from the site for study processes.

Grant their duly informed consent. Exclusion Criteria Subject lacking the mental capacity to understand the processes which imply their participation in the study and thus,not capable of granting their participation in a voluntary manner.

History of hypersensitivity to the medicines being studied. Daily intake of at least 240ml of grape juice or sporadic ingestion of 1 liter. Potentially fertile women without a safe family planning method, who wish to become pregnant during the study, are already pregnant or in lactation period.

Having on Globorisk scale for Mexicans, or as an associated risk factor, a high stratification for cardiovascular risk.

Basal laboratory values with elevation of ALT 1.5 times larger than the upper limit considered normal according to international units.

Basal laboratory values with elevation of CPK not attributable to physical activity.

Subjects who are under anti-coagulant treatment, suffer from coagulation disorders, or any circumstance which contraindicates the taking of a blood.

History of acute myocardial infarction, unstable angina, some confirmed coronopathy, arrhythmias, congestive cardiac failure or cerebrovascular disease.

History of muscular conditions of the genetic type or of rhabdomyolysis in patient or first degree relative.

History or diagnose of congenital hepatic disorders, chronic infection by hepatitis virus, hepatitis with fatty liver, alcoholic hepatitis, primary biliary cirrhosis, primary sclerosis, cholangitis or hepatic failure.

History or diagnose of congenital renal disorders, chronic renal failure, acute renal damage or nephritic syndrome.

History of infection by Human Immunodeficiency Virus. History of Acute or Chronic Pancreatitis. History of the following endocrine diseases: non-controlled Diabetes Mellitus, lipodystrophy, thyroid disorders, Cushing Syndrome and/or Polycystic Ovary Syndrome.

Diseases which compromise immunity such as Systemic Lupus Erythematous, Rheumatoid Arthritis, Antiphospholipid Antibodies Syndrome or Psoriasis.

Diseases by deposit such as Gaucher Disease, disease by glycogen deposit, Tay-Sachs juvenile disease or Niemann Pick Disease.

Diagnose of Kawasaki Disease, Werner Syndrome, intermittent acute Porphyria, Idiopathic Hyperkalemia or Klinefelter Syndrome.

Suffer from Idiopathic Hyperkalemia, Klinefelter Syndrome, Werner Syndrome, Kawasaki Disease or Porphyria.

History of epilepsy. History or diagnose of alcoholism. Intake of more than 20g of alcohol per day. User of marihuana. User of illegal drugs.

Intake of medicines with pharmacologic interaction which increase or decrease the efficacy of L-Carnitine and/or atorvastatin or alter the lipids in blood such as:

Macrolide antibiotics: Erythromycin, Telithromycin and Clarithromycin. Azole anti-fungi: Ketoconazole, Itraconazole, Fluconazole and Nefazodone. Quercetin, Amiodarone, Aprepitant, Cimetidine, Ciprofloxacin, Cyclosporine, Diltiazem, Imatinib, Echinacea, Enoxacin, Ergotamine, Metronidazole, Mifepristone, Tofisopam, Gestodene, Verapamil, Mibefradil, Fluoxetine, Phenobarbital, Carbamazepine, Phenytoin, Rifampin, Modafinil, Glucocorticoids, Felbamate, Rosiglitazone, Griseofulvin, Pioglitazone, Gemfibrozil, Clofibrate, Fenofibrate, Niacin, Nefazodone, Cholestyramine, Colchicine, Colestipol, Primidone, Topiramate, Troglitazone, Rifabutin, Digoxin, Thiazides, anabolic Steroids, Progestogens, Estrogens, Danazol, Amiodarone, fibric Acid, docosahexaenoic acid, Isotretinoine, Immunosuppressives, protease inhibitors of HIV or of the Hepatitis C Virus, Inhibitors of the co-transport of sodium-glucose, Tamoxifen, Raloxifene, non-selective Beta blockers, biliary acid sequestrants, asparginase, Sirolimus and Interferon.

Patients who have been diagnosed with terminal conditions. Patients with recent Cancer diagnose or undergoing any type of therapy for same. Patients who have suffered skin cancer not of the melanoma type and have been cured and haven't been on treatment for at least 1 year before the start of their participation in the study may enter.

Patients under lipid lowering treatment and who, because of their clinical condition aren't candidates to the period of lavage or detoxification; or well reject same.

Been participating in another clinical trial or having concluded their participation in the 30 days previous to beginning their participation in this study.

Any other which, at the Investigator's criteria, puts at risk the safety of the participant and/or interferes with the results of the study.

Medicine L-Carnitine, Atorvastatin Dose L-Carnitine 1 g + Atorvastatin 20 mg daily for 6 months and Atorvastatin 20 mg daily for 6 months

Efficacy criteria:

The efficacy of the combined treatment vs. atorvastatin in mono-therapy for dyslipidemia will be compared, through evaluation of the variability of the biochemical parameters at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Mexicans between 35 and 75 years of age.
* Gender indistinct.
* Patient with abnormal lipid profile considered as serum levels of Cholesterol LDL of 100mg/dl or greater, obtained by laboratory parameters.
* Not being under pharmacologic treatment to manage its dyslipidemia or accept to suspend current treatment and be evaluated for inclusion in the next 3 weeks starting on the day of initial evaluation.
* Women in fertile stage with a safe, hormonal-free family planning method. A safe planning method includes surgical methods in women, intrauterine device that doesn't release progestines and use of preservative in all their sexual relations.
* Women in fertile stage who don't wish to become pregnant during their participation in the study.
* Post-menopause women or with hysterectomy history.
* Have a fixed and/or mobile telephone and accept to receive calls from the site for study processes.
* Grant their duly informed consent.

Exclusion Criteria:

* Subject lacking the mental capacity to understand the processes which imply their participation in the study and thus, not capable of granting their participation in a voluntary manner
* History of hypersensitivity to the medicines being studied.
* Daily intake of at least 240 mL of grape juice or sporadic ingestion of 1 liter.
* Potentially fertile women without a safe family planning method, who wish to become pregnant during the study, are already pregnant or in lactation period.
* Having on Globorisk scale for Mexicans, or as an associated risk factor, a high stratification for cardiovascular risk.
* Basal laboratory values with elevation of ALT 1.5 times larger than the upper limit considered normal according to international units.

Basal laboratory values with elevation of CPK not attributable to physical activity.

* Subjects who are under anticoagulant treatment, suffer from coagulation disorders, or any circumstance which contraindicates the taking of a blood.
* History of acute myocardial infarction, unstable angina, some confirmed coronopathy, arrhythmias, congestive cardiac failure or cerebrovascular disease.
* History of muscular conditions of the genetic type or of rhabdomyolysis in the patient or first degree relative.
* History or diagnose of congenital hepatic disorders, chronic infection by hepatitis virus, hepatitis with fatty liver, alcoholic hepatitis, primary biliary cirrhosis, primary sclerosis, cholangitis or hepatic failure.
* History or diagnose of congenital renal disorders, chronic renal failure, acute renal damage or nephritic syndrome.
* History of infection by Human Immunodeficiency Virus.
* History of Acute or Chronic Pancreatitis.
* History of the following endocrine diseases: non controlled Diabetes Mellitus, lipodystrophy, thyroid disorders, Cushing Syndrome and or Polycystic Ovary Syndrome.
* Diseases which compromise immunity such as Systemic Lupus Erythematous, Rheumatoid Arthritis, Antiphospholipid Antibodies Syndrome or Psoriasis.

Diseases by deposit such as Gaucher Disease, disease by glycogen deposit, Tay Sachs juvenile disease or Niemann Pick Disease.

* Diagnose of Kawasaki Disease, Werner Syndrome, intermittent acute Porphyria, Idiopathic Hyperkalemia or Klinefelter Syndrome
* Suffer from Idiopathic Hyperkalemia, Klinefelter Syndrome, Werner Syndrome, Kawasaki Disease or Porphyria.
* History of epilepsy.
* History or diagnose of alcoholism.
* Intake of more than 20 grams of alcohol per day.
* User of marihuana.
* User of illegal drugs.
* Intake of medicines with pharmacologic interaction which increase or decrease the efficacy of L Carnitine and or atorvastatin or alter the lipids in blood such as Erythromycin, Telithromycin and Clarithromycin. Azole antifungi as Ketoconazole, Itraconazole, Fluconazole and Nefazodone. Quercetin, Amiodarone, Aprepitant, Cimetidine, Ciprofloxacin, Cyclosporine, Diltiazem, Imatinib, Echinacea, Enoxacin, Ergotamine, Metronidazole, Mifepristone, Tofisopam, Gestodene, Verapamil, Mibefradil, Fluoxetine, Phenobarbital, Carbamazepine, Phenytoin, Rifampin, Modafinil, Glucocorticoids, Felbamate, Rosiglitazone, Griseofulvin, Pioglitazone, Gemfibrozil, Clofibrate, Fenofibrate, Niacin, Nefazodone, Cholestyramine, Colchicine, Colestipol, Primidone, Topiramate, Troglitazone, Rifabutin, Digoxin, Thiazides, anabolic Steroids, Progestogens, Estrogens, Danazol, Amiodarone, fibric Acid, docosahexaenoic acid, Isotretinoine, Immunosuppressives, protease inhibitors of HIV or of the Hepatitis C Virus, Inhibitors of the cotransport of sodium glucose, Tamoxifen, Raloxifene, non selective Beta blockers, biliary acid sequestrants, asparginase, Sirolimus and Interferon.
* Patients who have been diagnosed with terminal conditions.
* Patients with recent Cancer diagnose or undergoing any type of therapy for same.
* Patients who have suffered skin cancer not of the melanoma type and have been cured and haven't been on treatment for at least 1 year before the start of their participation in the study may enter.
* Patients under lipid lowering treatment and who, because of their clinical condition aren't candidates to the period of lavage or detoxification; or well reject it.
* Being participating in another clinical trial or having concluded their participation in the 30 days previous to beginning their participation in this study.
* Any other which, at the Investigator's criteria, puts at risk the safety of the participant and or interferes with the results of the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of experimental treatment by the change in Cholesterol LDL | 6 months
  Evaluate the change of atorvastatin + l-carnitine vs. atorvastatin alone for dyslipidemia, through change of C-LDL in mg/dl

SECONDARY OUTCOMES:
Efficacy of experimental treatment by the change in Cholesterol no-HDL | 6 months
  Evaluate the change of Cholesterol no-HDL in Mexican adults with dyslipidemia through the use of oral route L-carnitine + atorvastatin in comparison with the use of Atorvastatin, after six months of treatment.
Efficacy of experimental treatment by the change in Total serum Cholesterol | 6 months
  Evaluate the change of serum levels of Cholesterol in mg/dl in Mexican adults with dyslipidemia through the use of oral route L-carnitine + atorvastatin in comparison with the use of Atorvastatin, after six months of treatment.
Efficacy of experimental treatment by the change in Triglycerides | 6 months
  Evaluate the reduction of serum levels of Triglycerides in mg/dl in Mexican adults with dyslipidemia through the use of oral route L-carnitine + atorvastatin in comparison with the use of Atorvastatin, after six months of treatment
Efficacy of experimental treatment by the change in Cholesterol HDL | 6 months
  Evaluate the change of serum levels of Cholesterol HDL in mg/dl in Mexican adults with dyslipidemia through the use of oral route L-carnitine + atorvastatin in comparison with the use of Atorvastatin, after six months of treatment
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | 6 months
  Evaluate the incidence, of serious and non-serious adverse events related through the oral route administration of L-carnitine + atorvastatin in comparison with the use of Atorvastatin, after six months of treatment in the subjects participating in the study

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Cruz Valdez, PhD, Principal Investigator — Instituto Nacional de Salud Pública; José Flores Figueroa, PhD, Principal Investigator — JM Research, SC
Locations (1):
- Laboratorios Grossman Sa, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bou Malham S, Goldberg AC. Cardiovascular risk reduction: the future of cholesterol lowering drugs. Curr Opin Pharmacol. 2016 Apr;27:62-9. doi: 10.1016/j.coph.2016.01.007. Epub 2016 Mar 2. PMID 26939026
- [Result] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Result] Rosenson RS, Baker SK, Jacobson TA, Kopecky SL, Parker BA, The National Lipid Association's Muscle Safety Expert Panel. An assessment by the Statin Muscle Safety Task Force: 2014 update. J Clin Lipidol. 2014 May-Jun;8(3 Suppl):S58-71. doi: 10.1016/j.jacl.2014.03.004. PMID 24793443
- [Result] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923
- [Result] Lee BJ, Lin JS, Lin YC, Lin PT. Effects of L-carnitine supplementation on lipid profiles in patients with coronary artery disease. Lipids Health Dis. 2016 Jun 17;15:107. doi: 10.1186/s12944-016-0277-5. PMID 27317162
- [Result] Chawla A, Repa JJ, Evans RM, Mangelsdorf DJ. Nuclear receptors and lipid physiology: opening the X-files. Science. 2001 Nov 30;294(5548):1866-70. doi: 10.1126/science.294.5548.1866. PMID 11729302
- [Result] Barter PJ, Rye KA. Relationship between the concentration and antiatherogenic activity of high-density lipoproteins. Curr Opin Lipidol. 2006 Aug;17(4):399-403. doi: 10.1097/01.mol.0000236365.40969.af. PMID 16832163
- [Result] Cooney MT, Dudina A, De Bacquer D, Wilhelmsen L, Sans S, Menotti A, De Backer G, Jousilahti P, Keil U, Thomsen T, Whincup P, Graham IM; SCORE investigators. HDL cholesterol protects against cardiovascular disease in both genders, at all ages and at all levels of risk. Atherosclerosis. 2009 Oct;206(2):611-6. doi: 10.1016/j.atherosclerosis.2009.02.041. Epub 2009 Mar 19. PMID 19375079
- [Result] Anderson TJ, Gregoire J, Hegele RA, Couture P, Mancini GB, McPherson R, Francis GA, Poirier P, Lau DC, Grover S, Genest J Jr, Carpentier AC, Dufour R, Gupta M, Ward R, Leiter LA, Lonn E, Ng DS, Pearson GJ, Yates GM, Stone JA, Ur E. 2012 update of the Canadian Cardiovascular Society guidelines for the diagnosis and treatment of dyslipidemia for the prevention of cardiovascular disease in the adult. Can J Cardiol. 2013 Feb;29(2):151-67. doi: 10.1016/j.cjca.2012.11.032. PMID 23351925
- [Result] Wadhera RK, Steen DL, Khan I, Giugliano RP, Foody JM. A review of low-density lipoprotein cholesterol, treatment strategies, and its impact on cardiovascular disease morbidity and mortality. J Clin Lipidol. 2016 May-Jun;10(3):472-89. doi: 10.1016/j.jacl.2015.11.010. Epub 2015 Nov 25. PMID 27206934
- [Result] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Result] Aguilar-Salinas CA, Canizales-Quinteros S, Rojas-Martinez R, Garcia-Garcia E, Olaiz-Fernandez G, Gomez-Perez FJ, Tusie-Luna MT. [Succesful collaborations between three Mexican institutions for research on dislipidemias, obesity and diabetes]. Gac Med Mex. 2007 Sep-Oct;143(5):355-64. Spanish. PMID 18246928
- [Result] Escobedo-de la Pena J, de Jesus-Perez R, Schargrodsky H, Champagne B. [Prevalence of dyslipidemias in Mexico city and Its relation to other cardiovascular risk factors. Results from the CARMELA study]. Gac Med Mex. 2014 Mar-Apr;150(2):128-36. Spanish. PMID 24603993
- [Result] Aguilar Salinas CA, Zamora M, Gomez-Diaz RA, Mehta R, Gomez Perez FJ, Rull JA. Familial combined hyperlipidemia: controversial aspects of its diagnosis and pathogenesis. Semin Vasc Med. 2004 May;4(2):203-9. doi: 10.1055/s-2004-835379. PMID 15478042
- [Result] Badzioch MD, Igo RP Jr, Gagnon F, Brunzell JD, Krauss RM, Motulsky AG, Wijsman EM, Jarvik GP. Low-density lipoprotein particle size loci in familial combined hyperlipidemia: evidence for multiple loci from a genome scan. Arterioscler Thromb Vasc Biol. 2004 Oct;24(10):1942-50. doi: 10.1161/01.ATV.0000143499.09575.93. Epub 2004 Aug 26. PMID 15331429
- [Result] Sniderman AD, Castro Cabezas M, Ribalta J, Carmena R, de Bruin TW, de Graaf J, Erkelens DW, Humphries SE, Masana L, Real JT, Talmud PJ, Taskinen MR. A proposal to redefine familial combined hyperlipidaemia -- third workshop on FCHL held in Barcelona from 3 to 5 May 2001, during the scientific sessions of the European Society for Clinical Investigation. Eur J Clin Invest. 2002 Feb;32(2):71-3. doi: 10.1046/j.1365-2362.2002.00941.x. No abstract available. PMID 11895451
- [Result] Veerkamp MJ, de Graaf J, Bredie SJ, Hendriks JC, Demacker PN, Stalenhoef AF. Diagnosis of familial combined hyperlipidemia based on lipid phenotype expression in 32 families: results of a 5-year follow-up study. Arterioscler Thromb Vasc Biol. 2002 Feb 1;22(2):274-82. doi: 10.1161/hq0202.104059. PMID 11834528
- [Result] Sullivan DR, Hamilton-Craig I, van Bockxmeer F, Watts GF; CSANZ Cardiac Genetics Diseases Council Writing Group. INTERIM guidelines for the diagnosis and management of familial hypercholesterolaemia. Heart Lung Circ. 2012 Mar;21(3):159-62. doi: 10.1016/j.hlc.2011.11.006. Epub 2012 Jan 30. No abstract available. PMID 22364837
- [Result] Alonso R, Castillo S, Civeira F, Puzo J, de la Cruz JJ, Pocovi M, Mata P. [Heterozygous familial hypercholesterolemia in Spain. Description of 819 non related cases]. Med Clin (Barc). 2002 Apr 13;118(13):487-92. doi: 10.1016/s0025-7753(02)72428-7. Spanish. PMID 11975885
- [Result] Blom DJ, O'Neill FH, Marais AD. Screening for dysbetalipoproteinemia by plasma cholesterol and apolipoprotein B concentrations. Clin Chem. 2005 May;51(5):904-7. doi: 10.1373/clinchem.2004.047001. No abstract available. PMID 15855667
- [Result] Cohen JC, Boerwinkle E, Mosley TH Jr, Hobbs HH. Sequence variations in PCSK9, low LDL, and protection against coronary heart disease. N Engl J Med. 2006 Mar 23;354(12):1264-72. doi: 10.1056/NEJMoa054013. PMID 16554528
- [Result] Abifadel M, Varret M, Rabes JP, Allard D, Ouguerram K, Devillers M, Cruaud C, Benjannet S, Wickham L, Erlich D, Derre A, Villeger L, Farnier M, Beucler I, Bruckert E, Chambaz J, Chanu B, Lecerf JM, Luc G, Moulin P, Weissenbach J, Prat A, Krempf M, Junien C, Seidah NG, Boileau C. Mutations in PCSK9 cause autosomal dominant hypercholesterolemia. Nat Genet. 2003 Jun;34(2):154-6. doi: 10.1038/ng1161. PMID 12730697
- [Result] Garcia CK, Wilund K, Arca M, Zuliani G, Fellin R, Maioli M, Calandra S, Bertolini S, Cossu F, Grishin N, Barnes R, Cohen JC, Hobbs HH. Autosomal recessive hypercholesterolemia caused by mutations in a putative LDL receptor adaptor protein. Science. 2001 May 18;292(5520):1394-8. doi: 10.1126/science.1060458. Epub 2001 Apr 26. PMID 11326085
- [Result] Vodnala D, Rubenfire M, Brook RD. Secondary causes of dyslipidemia. Am J Cardiol. 2012 Sep 15;110(6):823-5. doi: 10.1016/j.amjcard.2012.04.062. Epub 2012 Jun 2. PMID 22658245
- [Result] Vaziri ND. Disorders of lipid metabolism in nephrotic syndrome: mechanisms and consequences. Kidney Int. 2016 Jul;90(1):41-52. doi: 10.1016/j.kint.2016.02.026. Epub 2016 Apr 26. PMID 27165836
- [Result] de Jager DJ, Grootendorst DC, Jager KJ, van Dijk PC, Tomas LM, Ansell D, Collart F, Finne P, Heaf JG, De Meester J, Wetzels JF, Rosendaal FR, Dekker FW. Cardiovascular and noncardiovascular mortality among patients starting dialysis. JAMA. 2009 Oct 28;302(16):1782-9. doi: 10.1001/jama.2009.1488. PMID 19861670
- [Result] Glass TR, Ungsedhapand C, Wolbers M, Weber R, Vernazza PL, Rickenbach M, Furrer H, Bernasconi E, Cavassini M, Hirschel B, Battegay M, Bucher HC; Swiss HIV Cohort Study. Prevalence of risk factors for cardiovascular disease in HIV-infected patients over time: the Swiss HIV Cohort Study. HIV Med. 2006 Sep;7(6):404-10. doi: 10.1111/j.1468-1293.2006.00400.x. PMID 16903986
- [Result] Reiner Z, Catapano AL, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs RH, Kjekshus JK, Perrone Filardi P, Riccardi G, Storey RF, David W; Clinical Practice Guidelines Committee of the Spanish Society of Cardiology. [ESC/EAS Guidelines for the management of dyslipidaemias]. Rev Esp Cardiol. 2011 Dec;64(12):1168.e1-1168.e60. doi: 10.1016/j.recesp.2011.09.014. No abstract available. Spanish. PMID 22115524
- [Result] Bays HE, Jones PH, Orringer CE, Brown WV, Jacobson TA. National Lipid Association Annual Summary of Clinical Lipidology 2016. J Clin Lipidol. 2016 Jan-Feb;10(1 Suppl):S1-43. doi: 10.1016/j.jacl.2015.08.002. PMID 26891998
- [Result] Levenson JW, Skerrett PJ, Gaziano JM. Reducing the global burden of cardiovascular disease: the role of risk factors. Prev Cardiol. 2002 Fall;5(4):188-99. doi: 10.1111/j.1520-037x.2002.00564.x. PMID 12417828
- [Result] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB Sr, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PWF. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2935-2959. doi: 10.1016/j.jacc.2013.11.005. Epub 2013 Nov 12. No abstract available. PMID 24239921
- [Result] Austin MA, McKnight B, Edwards KL, Bradley CM, McNeely MJ, Psaty BM, Brunzell JD, Motulsky AG. Cardiovascular disease mortality in familial forms of hypertriglyceridemia: A 20-year prospective study. Circulation. 2000 Jun 20;101(24):2777-82. doi: 10.1161/01.cir.101.24.2777. PMID 10859281
- [Result] Blair HC, Sepulveda J, Papachristou DJ. Nature and nurture in atherosclerosis: The roles of acylcarnitine and cell membrane-fatty acid intermediates. Vascul Pharmacol. 2016 Mar;78:17-23. doi: 10.1016/j.vph.2015.06.012. Epub 2015 Jun 30. PMID 26133667
- [Result] Stamler J, Neaton JD. The Multiple Risk Factor Intervention Trial (MRFIT)--importance then and now. JAMA. 2008 Sep 17;300(11):1343-5. doi: 10.1001/jama.300.11.1343. No abstract available. PMID 18799447
- [Result] Acosta-Cazares B, Escobedo-de la Pena J. High burden of cardiovascular disease risk factors in Mexico: An epidemic of ischemic heart disease that may be on its way? Am Heart J. 2010 Aug;160(2):230-6. doi: 10.1016/j.ahj.2010.05.016. PMID 20691826
- [Result] Schaefer EJ, Levy RI. Pathogenesis and management of lipoprotein disorders. N Engl J Med. 1985 May 16;312(20):1300-10. doi: 10.1056/NEJM198505163122007. No abstract available. PMID 3887163
- [Result] Lloyd-Jones DM, Leip EP, Larson MG, D'Agostino RB, Beiser A, Wilson PW, Wolf PA, Levy D. Prediction of lifetime risk for cardiovascular disease by risk factor burden at 50 years of age. Circulation. 2006 Feb 14;113(6):791-8. doi: 10.1161/CIRCULATIONAHA.105.548206. Epub 2006 Feb 6. PMID 16461820
- [Result] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Result] Hajifathalian K, Ueda P, Lu Y, Woodward M, Ahmadvand A, Aguilar-Salinas CA, Azizi F, Cifkova R, Di Cesare M, Eriksen L, Farzadfar F, Ikeda N, Khalili D, Khang YH, Lanska V, Leon-Munoz L, Magliano D, Msyamboza KP, Oh K, Rodriguez-Artalejo F, Rojas-Martinez R, Shaw JE, Stevens GA, Tolstrup J, Zhou B, Salomon JA, Ezzati M, Danaei G. A novel risk score to predict cardiovascular disease risk in national populations (Globorisk): a pooled analysis of prospective cohorts and health examination surveys. Lancet Diabetes Endocrinol. 2015 May;3(5):339-55. doi: 10.1016/S2213-8587(15)00081-9. Epub 2015 Mar 26. PMID 25819778
- [Result] Bays HE. A lipidologist perspective of global lipid guidelines and recommendations, part 2: Lipid treatment goals. J Clin Lipidol. 2016 Mar-Apr;10(2):240-64. doi: 10.1016/j.jacl.2015.11.006. Epub 2015 Dec 2. PMID 27055955
- [Result] Bouhairie VE, Goldberg AC. Familial Hypercholesterolemia. Endocrinol Metab Clin North Am. 2016 Mar;45(1):1-16. doi: 10.1016/j.ecl.2015.09.001. PMID 26892994
- [Result] Hopkins PN, Toth PP, Ballantyne CM, Rader DJ; National Lipid Association Expert Panel on Familial Hypercholesterolemia. Familial hypercholesterolemias: prevalence, genetics, diagnosis and screening recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Clin Lipidol. 2011 Jun;5(3 Suppl):S9-17. doi: 10.1016/j.jacl.2011.03.452. Epub 2011 Apr 3. No abstract available. PMID 21600530
- [Result] Miller M, Cannon CP, Murphy SA, Qin J, Ray KK, Braunwald E; PROVE IT-TIMI 22 Investigators. Impact of triglyceride levels beyond low-density lipoprotein cholesterol after acute coronary syndrome in the PROVE IT-TIMI 22 trial. J Am Coll Cardiol. 2008 Feb 19;51(7):724-30. doi: 10.1016/j.jacc.2007.10.038. PMID 18279736
- [Result] Zhao D, Liu J, Xie W, Qi Y. Cardiovascular risk assessment: a global perspective. Nat Rev Cardiol. 2015 May;12(5):301-11. doi: 10.1038/nrcardio.2015.28. Epub 2015 Mar 10. PMID 25754885
- [Result] Sheridan SL, Viera AJ, Krantz MJ, Ice CL, Steinman LE, Peters KE, Kopin LA, Lungelow D; Cardiovascular Health Intervention Research and Translation Network Work Group on Global Coronary Heart Disease Risk. The effect of giving global coronary risk information to adults: a systematic review. Arch Intern Med. 2010 Feb 8;170(3):230-9. doi: 10.1001/archinternmed.2009.516. PMID 20142567
- [Result] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Result] Kraus WE, Houmard JA, Duscha BD, Knetzger KJ, Wharton MB, McCartney JS, Bales CW, Henes S, Samsa GP, Otvos JD, Kulkarni KR, Slentz CA. Effects of the amount and intensity of exercise on plasma lipoproteins. N Engl J Med. 2002 Nov 7;347(19):1483-92. doi: 10.1056/NEJMoa020194. PMID 12421890
- [Result] Lozano P, Henrikson NB, Morrison CC, Dunn J, Nguyen M, Blasi PR, Whitlock EP. Lipid Screening in Childhood and Adolescence for Detection of Multifactorial Dyslipidemia: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2016 Aug 9;316(6):634-44. doi: 10.1001/jama.2016.6423. PMID 27532918
- [Result] Avis HJ, Vissers MN, Stein EA, Wijburg FA, Trip MD, Kastelein JJ, Hutten BA. A systematic review and meta-analysis of statin therapy in children with familial hypercholesterolemia. Arterioscler Thromb Vasc Biol. 2007 Aug;27(8):1803-10. doi: 10.1161/ATVBAHA.107.145151. Epub 2007 Jun 14. PMID 17569881
- [Result] Robinson JG, Wang S, Jacobson TA. Meta-analysis of comparison of effectiveness of lowering apolipoprotein B versus low-density lipoprotein cholesterol and nonhigh-density lipoprotein cholesterol for cardiovascular risk reduction in randomized trials. Am J Cardiol. 2012 Nov 15;110(10):1468-76. doi: 10.1016/j.amjcard.2012.07.007. Epub 2012 Aug 17. PMID 22906895
- [Result] Bays H, Cohen DE, Chalasani N, Harrison SA, The National Lipid Association's Statin Safety Task Force. An assessment by the Statin Liver Safety Task Force: 2014 update. J Clin Lipidol. 2014 May-Jun;8(3 Suppl):S47-57. doi: 10.1016/j.jacl.2014.02.011. PMID 24793441
- [Result] American Diabetes Association. (8) Cardiovascular disease and risk management. Diabetes Care. 2015 Jan;38 Suppl:S49-57. doi: 10.2337/dc15-S011. No abstract available. PMID 25537708
- [Result] Jacobson TA, Maki KC, Orringer CE, Jones PH, Kris-Etherton P, Sikand G, La Forge R, Daniels SR, Wilson DP, Morris PB, Wild RA, Grundy SM, Daviglus M, Ferdinand KC, Vijayaraghavan K, Deedwania PC, Aberg JA, Liao KP, McKenney JM, Ross JL, Braun LT, Ito MK, Bays HE, Brown WV, Underberg JA; NLA Expert Panel. National Lipid Association Recommendations for Patient-Centered Management of Dyslipidemia: Part 2. J Clin Lipidol. 2015 Nov-Dec;9(6 Suppl):S1-122.e1. doi: 10.1016/j.jacl.2015.09.002. Epub 2015 Sep 18. PMID 26699442
- [Result] Ble A, Hughes PM, Delgado J, Masoli JA, Bowman K, Zirk-Sadowski J, Mujica Mota RE, Henley WE, Melzer D. Safety and Effectiveness of Statins for Prevention of Recurrent Myocardial Infarction in 12 156 Typical Older Patients: A Quasi-Experimental Study. J Gerontol A Biol Sci Med Sci. 2017 Feb;72(2):243-250. doi: 10.1093/gerona/glw082. Epub 2016 May 4. PMID 27146371
- [Result] Writing Committee; Lloyd-Jones DM, Morris PB, Ballantyne CM, Birtcher KK, Daly DD Jr, DePalma SM, Minissian MB, Orringer CE, Smith SC Jr. 2016 ACC Expert Consensus Decision Pathway on the Role of Non-Statin Therapies for LDL-Cholesterol Lowering in the Management of Atherosclerotic Cardiovascular Disease Risk: A Report of the American College of Cardiology Task Force on Clinical Expert Consensus Documents. J Am Coll Cardiol. 2016 Jul 5;68(1):92-125. doi: 10.1016/j.jacc.2016.03.519. Epub 2016 Apr 1. No abstract available. PMID 27046161
- [Result] Kellick KA, Bottorff M, Toth PP, The National Lipid Association's Safety Task Force. A clinician's guide to statin drug-drug interactions. J Clin Lipidol. 2014 May-Jun;8(3 Suppl):S30-46. doi: 10.1016/j.jacl.2014.02.010. PMID 24793440
- [Result] Paiva H, Thelen KM, Van Coster R, Smet J, De Paepe B, Mattila KM, Laakso J, Lehtimaki T, von Bergmann K, Lutjohann D, Laaksonen R. High-dose statins and skeletal muscle metabolism in humans: a randomized, controlled trial. Clin Pharmacol Ther. 2005 Jul;78(1):60-8. doi: 10.1016/j.clpt.2005.03.006. PMID 16003294
- [Result] Parker BA, Capizzi JA, Grimaldi AS, Clarkson PM, Cole SM, Keadle J, Chipkin S, Pescatello LS, Simpson K, White CM, Thompson PD. Effect of statins on skeletal muscle function. Circulation. 2013 Jan 1;127(1):96-103. doi: 10.1161/CIRCULATIONAHA.112.136101. Epub 2012 Nov 26. PMID 23183941
- [Result] Apostolopoulou M, Corsini A, Roden M. The role of mitochondria in statin-induced myopathy. Eur J Clin Invest. 2015 Jul;45(7):745-54. doi: 10.1111/eci.12461. Epub 2015 Jun 15. PMID 25991405
- [Result] Sattar N, Preiss D, Murray HM, Welsh P, Buckley BM, de Craen AJ, Seshasai SR, McMurray JJ, Freeman DJ, Jukema JW, Macfarlane PW, Packard CJ, Stott DJ, Westendorp RG, Shepherd J, Davis BR, Pressel SL, Marchioli R, Marfisi RM, Maggioni AP, Tavazzi L, Tognoni G, Kjekshus J, Pedersen TR, Cook TJ, Gotto AM, Clearfield MB, Downs JR, Nakamura H, Ohashi Y, Mizuno K, Ray KK, Ford I. Statins and risk of incident diabetes: a collaborative meta-analysis of randomised statin trials. Lancet. 2010 Feb 27;375(9716):735-42. doi: 10.1016/S0140-6736(09)61965-6. Epub 2010 Feb 16. PMID 20167359
- [Result] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Result] Ross S, D'Mello M, Anand SS, Eikelboom J; CARDIoGRAMplusC4D Consortium; Stewart AF, Samani NJ, Roberts R, Pare G. Effect of Bile Acid Sequestrants on the Risk of Cardiovascular Events: A Mendelian Randomization Analysis. Circ Cardiovasc Genet. 2015 Aug;8(4):618-27. doi: 10.1161/CIRCGENETICS.114.000952. Epub 2015 Jun 4. PMID 26043746
- [Result] Schoonjans K, Staels B, Auwerx J. Role of the peroxisome proliferator-activated receptor (PPAR) in mediating the effects of fibrates and fatty acids on gene expression. J Lipid Res. 1996 May;37(5):907-25. PMID 8725145
- [Result] Stanulovic V, Deric M, Popovic J. [Clinical trials of statins and fibrates --a meta-analysis]. Med Pregl. 2006 May-Jun;59(5-6):213-8. doi: 10.2298/mpns0606213s. Serbian. PMID 17039901
- [Result] Navarese EP, Kolodziejczak M, Schulze V, Gurbel PA, Tantry U, Lin Y, Brockmeyer M, Kandzari DE, Kubica JM, D'Agostino RB Sr, Kubica J, Volpe M, Agewall S, Kereiakes DJ, Kelm M. Effects of Proprotein Convertase Subtilisin/Kexin Type 9 Antibodies in Adults With Hypercholesterolemia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Jul 7;163(1):40-51. doi: 10.7326/M14-2957. PMID 25915661
- [Result] Brass EP. Supplemental carnitine and exercise. Am J Clin Nutr. 2000 Aug;72(2 Suppl):618S-23S. doi: 10.1093/ajcn/72.2.618S. PMID 10919968
- [Result] Serban MC, Sahebkar A, Mikhailidis DP, Toth PP, Jones SR, Muntner P, Blaha MJ, Andrica F, Martin SS, Borza C, Lip GY, Ray KK, Rysz J, Hazen SL, Banach M. Impact of L-carnitine on plasma lipoprotein(a) concentrations: A systematic review and meta-analysis of randomized controlled trials. Sci Rep. 2016 Jan 12;6:19188. doi: 10.1038/srep19188. PMID 26754058
- [Result] Naini AE, Sadeghi M, Mortazavi M, Moghadasi M, Harandi AA. Oral carnitine supplementation for dyslipidemia in chronic hemodialysis patients. Saudi J Kidney Dis Transpl. 2012 May;23(3):484-8. PMID 22569432
- [Result] Emami Naini A, Moradi M, Mortazavi M, Amini Harandi A, Hadizadeh M, Shirani F, Basir Ghafoori H, Emami Naini P. Effects of Oral L-Carnitine Supplementation on Lipid Profile, Anemia, and Quality of Life in Chronic Renal Disease Patients under Hemodialysis: A Randomized, Double-Blinded, Placebo-Controlled Trial. J Nutr Metab. 2012;2012:510483. doi: 10.1155/2012/510483. Epub 2012 Jun 5. PMID 22720143
- [Result] Ferrari R, Merli E, Cicchitelli G, Mele D, Fucili A, Ceconi C. Therapeutic effects of L-carnitine and propionyl-L-carnitine on cardiovascular diseases: a review. Ann N Y Acad Sci. 2004 Nov;1033:79-91. doi: 10.1196/annals.1320.007. PMID 15591005
- [Result] Tiwari A, Bansal V, Chugh A, Mookhtiar K. Statins and myotoxicity: a therapeutic limitation. Expert Opin Drug Saf. 2006 Sep;5(5):651-66. doi: 10.1517/14740338.5.5.651. PMID 16907655
- [Result] Anfossi G, Massucco P, Bonomo K, Trovati M. Prescription of statins to dyslipidemic patients affected by liver diseases: a subtle balance between risks and benefits. Nutr Metab Cardiovasc Dis. 2004 Aug;14(4):215-24. doi: 10.1016/s0939-4753(04)80008-5. PMID 15553600
- [Result] Chatzizisis YS, Koskinas KC, Misirli G, Vaklavas C, Hatzitolios A, Giannoglou GD. Risk factors and drug interactions predisposing to statin-induced myopathy: implications for risk assessment, prevention and treatment. Drug Saf. 2010 Mar 1;33(3):171-87. doi: 10.2165/11319380-000000000-00000. PMID 20158283
- [Result] Arora R, Liebo M, Maldonado F. Statin-induced myopathy: the two faces of Janus. J Cardiovasc Pharmacol Ther. 2006 Jun;11(2):105-12. doi: 10.1177/1074248406288758. PMID 16891287
- [Result] Owczarek J, Jasinska M, Orszulak-Michalak D. Drug-induced myopathies. An overview of the possible mechanisms. Pharmacol Rep. 2005 Jan-Feb;57(1):23-34. PMID 15849374
- [Result] Armitage J. The safety of statins in clinical practice. Lancet. 2007 Nov 24;370(9601):1781-90. doi: 10.1016/S0140-6736(07)60716-8. PMID 17559928
- [Result] Law MR, Wald NJ, Rudnicka AR. Quantifying effect of statins on low density lipoprotein cholesterol, ischaemic heart disease, and stroke: systematic review and meta-analysis. BMJ. 2003 Jun 28;326(7404):1423. doi: 10.1136/bmj.326.7404.1423. PMID 12829554
- [Result] Arca M. Atorvastatin: a safety and tolerability profile. Drugs. 2007;67 Suppl 1:63-9. doi: 10.2165/00003495-200767001-00007. PMID 17910522
- [Result] Sever PS, Dahlof B, Poulter NR, Wedel H, Beevers G, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT investigators. Prevention of coronary and stroke events with atorvastatin in hypertensive patients who have average or lower-than-average cholesterol concentrations, in the Anglo-Scandinavian Cardiac Outcomes Trial--Lipid Lowering Arm (ASCOT-LLA): a multicentre randomised controlled trial. Lancet. 2003 Apr 5;361(9364):1149-58. doi: 10.1016/S0140-6736(03)12948-0. PMID 12686036
- [Result] Schwartz GG, Olsson AG, Ezekowitz MD, Ganz P, Oliver MF, Waters D, Zeiher A, Chaitman BR, Leslie S, Stern T; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Effects of atorvastatin on early recurrent ischemic events in acute coronary syndromes: the MIRACL study: a randomized controlled trial. JAMA. 2001 Apr 4;285(13):1711-8. doi: 10.1001/jama.285.13.1711. PMID 11277825
- [Result] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Result] LaRosa JC, Grundy SM, Waters DD, Shear C, Barter P, Fruchart JC, Gotto AM, Greten H, Kastelein JJ, Shepherd J, Wenger NK; Treating to New Targets (TNT) Investigators. Intensive lipid lowering with atorvastatin in patients with stable coronary disease. N Engl J Med. 2005 Apr 7;352(14):1425-35. doi: 10.1056/NEJMoa050461. Epub 2005 Mar 8. PMID 15755765
- [Result] Escobar C, Echarri R, Barrios V. Relative safety profiles of high dose statin regimens. Vasc Health Risk Manag. 2008;4(3):525-33. doi: 10.2147/vhrm.s2048. PMID 18827903
- [Result] Newman CB, Palmer G, Silbershatz H, Szarek M. Safety of atorvastatin derived from analysis of 44 completed trials in 9,416 patients. Am J Cardiol. 2003 Sep 15;92(6):670-6. doi: 10.1016/s0002-9149(03)00820-8. PMID 12972104
- [Result] Newman C, Tsai J, Szarek M, Luo D, Gibson E. Comparative safety of atorvastatin 80 mg versus 10 mg derived from analysis of 49 completed trials in 14,236 patients. Am J Cardiol. 2006 Jan 1;97(1):61-7. doi: 10.1016/j.amjcard.2005.07.108. Epub 2005 Nov 15. PMID 16377285
- [Result] Athyros VG, Papageorgiou AA, Symeonidis AN, Didangelos TP, Pehlivanidis AN, Bouloukos VI, Mikhailidis DP; GREACE Study Collaborative Group. Early benefit from structured care with atorvastatin in patients with coronary heart disease and diabetes mellitus. Angiology. 2003 Nov-Dec;54(6):679-90. doi: 10.1177/000331970305400607. PMID 14666956
- [Result] Patel SS, Kimmel PL, Singh A. New clinical practice guidelines for chronic kidney disease: a framework for K/DOQI. Semin Nephrol. 2002 Nov;22(6):449-58. doi: 10.1053/snep.2002.35973. PMID 12430089
- [Result] Wanner C, Krane V, Marz W, Olschewski M, Mann JF, Ruf G, Ritz E; German Diabetes and Dialysis Study Investigators. Atorvastatin in patients with type 2 diabetes mellitus undergoing hemodialysis. N Engl J Med. 2005 Jul 21;353(3):238-48. doi: 10.1056/NEJMoa043545. PMID 16034009
- [Result] Carter AL, Abney TO, Lapp DF. Biosynthesis and metabolism of carnitine. J Child Neurol. 1995 Nov;10 Suppl 2:S3-7. PMID 8576566
- [Result] Lee MS, Lee HJ, Lee HS, Kim Y. L-carnitine stimulates lipolysis via induction of the lipolytic gene expression and suppression of the adipogenic gene expression in 3T3-L1 adipocytes. J Med Food. 2006 Winter;9(4):468-73. doi: 10.1089/jmf.2006.9.468. PMID 17201631
- [Result] Stephens FB, Constantin-Teodosiu D, Laithwaite D, Simpson EJ, Greenhaff PL. A threshold exists for the stimulatory effect of insulin on plasma L-carnitine clearance in humans. Am J Physiol Endocrinol Metab. 2007 Feb;292(2):E637-41. doi: 10.1152/ajpendo.00508.2006. Epub 2006 Oct 17. PMID 17047160
- [Result] Rajasekar P, Anuradha CV. Effect of L-carnitine on skeletal muscle lipids and oxidative stress in rats fed high-fructose diet. Exp Diabetes Res. 2007;2007:72741. doi: 10.1155/2007/72741. PMID 17641743
- [Result] Evans AM, Fornasini G. Pharmacokinetics of L-carnitine. Clin Pharmacokinet. 2003;42(11):941-67. doi: 10.2165/00003088-200342110-00002. PMID 12908852
- [Result] Irat AM, Aktan F, Ozansoy G. Effects of L-carnitine treatment on oxidant/antioxidant state and vascular reactivity of streptozotocin-diabetic rat aorta. J Pharm Pharmacol. 2003 Oct;55(10):1389-95. doi: 10.1211/0022357021909. PMID 14607021
- [Result] Sayed-Ahmed MM, Khattab MM, Gad MZ, Mostafa N. L-carnitine prevents the progression of atherosclerotic lesions in hypercholesterolaemic rabbits. Pharmacol Res. 2001 Sep;44(3):235-42. doi: 10.1006/phrs.2001.0852. PMID 11529691
- [Result] Derosa G, Cicero AF, Gaddi A, Mugellini A, Ciccarelli L, Fogari R. The effect of L-carnitine on plasma lipoprotein(a) levels in hypercholesterolemic patients with type 2 diabetes mellitus. Clin Ther. 2003 May;25(5):1429-39. doi: 10.1016/s0149-2918(03)80130-3. PMID 12867219
- [Result] Bartel LL, Hussey JL, Shrago E. Perturbation of serum carnitine levels in human adults by chronic renal disease and dialysis therapy. Am J Clin Nutr. 1981 Jul;34(7):1314-20. doi: 10.1093/ajcn/34.7.1314. PMID 7258121
- [Result] Abdoli N, Azarmi Y, Eghbal MA. Mitigation of statins-induced cytotoxicity and mitochondrial dysfunction by L-carnitine in freshly-isolated rat hepatocytes. Res Pharm Sci. 2015 Mar-Apr;10(2):143-51. PMID 26487891
- [Result] DiNicolantonio JJ. CoQ10 and L-carnitine for statin myalgia? Expert Rev Cardiovasc Ther. 2012 Oct;10(10):1329-33. doi: 10.1586/erc.12.92. PMID 23190071
- [Result] Galvano F, Li Volti G, Malaguarnera M, Avitabile T, Antic T, Vacante M, Malaguarnera M. Effects of simvastatin and carnitine versus simvastatin on lipoprotein(a) and apoprotein(a) in type 2 diabetes mellitus. Expert Opin Pharmacother. 2009 Aug;10(12):1875-82. doi: 10.1517/14656560903081745. PMID 19618992
- [Result] Malaguarnera M, Vacante M, Motta M, Malaguarnera M, Li Volti G, Galvano F. Effect of L-carnitine on the size of low-density lipoprotein particles in type 2 diabetes mellitus patients treated with simvastatin. Metabolism. 2009 Nov;58(11):1618-23. doi: 10.1016/j.metabol.2009.05.014. Epub 2009 Jul 15. PMID 19604523
- [Result] Solfrizzi V, Capurso C, Colacicco AM, D'Introno A, Fontana C, Capurso SA, Torres F, Gadaleta AM, Koverech A, Capurso A, Panza F. Efficacy and tolerability of combined treatment with L-carnitine and simvastatin in lowering lipoprotein(a) serum levels in patients with type 2 diabetes mellitus. Atherosclerosis. 2006 Oct;188(2):455-61. doi: 10.1016/j.atherosclerosis.2005.11.024. Epub 2005 Dec 27. PMID 16384561
- [Result] Shojaei M, Djalali M, Khatami M, Siassi F, Eshraghian M. Effects of carnitine and coenzyme Q10 on lipid profile and serum levels of lipoprotein(a) in maintenance hemodialysis patients on statin therapy. Iran J Kidney Dis. 2011 Mar;5(2):114-8. PMID 21368390
- [Result] Rtveladze K, Marsh T, Barquera S, Sanchez Romero LM, Levy D, Melendez G, Webber L, Kilpi F, McPherson K, Brown M. Obesity prevalence in Mexico: impact on health and economic burden. Public Health Nutr. 2014 Jan;17(1):233-9. doi: 10.1017/S1368980013000086. Epub 2013 Feb 1. PMID 23369462
- [Result] Viera AJ, Sheridan SL. Global risk of coronary heart disease: assessment and application. Am Fam Physician. 2010 Aug 1;82(3):265-74. PMID 20672791
- [Result] Ajufo E, Rader DJ. Recent advances in the pharmacological management of hypercholesterolaemia. Lancet Diabetes Endocrinol. 2016 May;4(5):436-46. doi: 10.1016/S2213-8587(16)00074-7. Epub 2016 Mar 21. PMID 27012540
- [Result] Collins R, Reith C, Emberson J, Armitage J, Baigent C, Blackwell L, Blumenthal R, Danesh J, Smith GD, DeMets D, Evans S, Law M, MacMahon S, Martin S, Neal B, Poulter N, Preiss D, Ridker P, Roberts I, Rodgers A, Sandercock P, Schulz K, Sever P, Simes J, Smeeth L, Wald N, Yusuf S, Peto R. Interpretation of the evidence for the efficacy and safety of statin therapy. Lancet. 2016 Nov 19;388(10059):2532-2561. doi: 10.1016/S0140-6736(16)31357-5. Epub 2016 Sep 8. PMID 27616593
- [Result] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Result] Rosas-Peralta M, Santos-Martinez LE, Magana-Serrano JA, Valencia-Sanchez JS, Garrido-Garduno M, Perez-Rodriguez G. [Methodology for superiority versus equivalence and non-inferior clinical studies. A practical review]. Rev Med Inst Mex Seguro Soc. 2016 May-Jun;54(3):344-53. Spanish. PMID 27100981
- [Result] De Vivo DC, Bohan TP, Coulter DL, Dreifuss FE, Greenwood RS, Nordli DR Jr, Shields WD, Stafstrom CE, Tein I. L-carnitine supplementation in childhood epilepsy: current perspectives. Epilepsia. 1998 Nov;39(11):1216-25. doi: 10.1111/j.1528-1157.1998.tb01315.x. PMID 9821988
- [Result] Van Oudheusden LJ, Scholte HR. Efficacy of carnitine in the treatment of children with attention-deficit hyperactivity disorder. Prostaglandins Leukot Essent Fatty Acids. 2002 Jul;67(1):33-8. doi: 10.1054/plef.2002.0378. PMID 12213433
- [Result] Rizos I. Three-year survival of patients with heart failure caused by dilated cardiomyopathy and L-carnitine administration. Am Heart J. 2000 Feb;139(2 Pt 3):S120-3. doi: 10.1067/mhj.2000.103917. PMID 10650325
- [Result] Ellaway C, Williams K, Leonard H, Higgins G, Wilcken B, Christodoulou J. Rett syndrome: randomized controlled trial of L-carnitine. J Child Neurol. 1999 Mar;14(3):162-7. doi: 10.1177/088307389901400306. PMID 10190267
- [Result] Plioplys AV, Plioplys S. Amantadine and L-carnitine treatment of Chronic Fatigue Syndrome. Neuropsychobiology. 1997;35(1):16-23. doi: 10.1159/000119325. PMID 9018019
- [Result] Campos Y, Huertas R, Lorenzo G, Bautista J, Gutierrez E, Aparicio M, Alesso L, Arenas J. Plasma carnitine insufficiency and effectiveness of L-carnitine therapy in patients with mitochondrial myopathy. Muscle Nerve. 1993 Feb;16(2):150-3. doi: 10.1002/mus.880160205. PMID 8429838
- [Result] Cherchi A, Lai C, Angelino F, Trucco G, Caponnetto S, Mereto PE, Rosolen G, Manzoli U, Schiavoni G, Reale A, et al. Effects of L-carnitine on exercise tolerance in chronic stable angina: a multicenter, double-blind, randomized, placebo controlled crossover study. Int J Clin Pharmacol Ther Toxicol. 1985 Oct;23(10):569-72. PMID 3905631
- [Result] Harper P, Elwin CE, Cederblad G. Pharmacokinetics of intravenous and oral bolus doses of L-carnitine in healthy subjects. Eur J Clin Pharmacol. 1988;35(5):555-62. doi: 10.1007/BF00558253. PMID 3234464
- See also: World Health Organization: Global Status report on non-communicable diseases 2014. — http://who.int
- See also: Protocolo clínico para el diagnóstico y tratamiento de las Dislipidemias. CENAPRECE, Secretaría e Salud, D.F. México. — http://www.cenaprece.salud.gob.mx/
- See also: Treatment of lipids (including hypercholesterolemia) in secondary prevention. — http://www.uptodate.com.
- See also: Organization for Economic Cooperation and Development. — http://www.oecd.org/health/

DOCUMENTS (1):
  • Study Protocol (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03696940/Prot_000.pdf